CLINICAL TRIAL: NCT06669221
Title: Effectiveness of Early Intervention in Transfusion Independent Aplastic Anemia: a Retrospective Medical Claims Database Study
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CETB115EJP05
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Aplastic Anemia (AA)
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Early drug intervention group: Patients who had at least one prescription record associated with any of the drug treatments of interest (cyclosporine A, eltrombopag, romiplostin, danazol, or methenolone) during each period of interest before the first transfusion record during the follow-up period.
- Watchful observation group: Patients with no prescription record associated with any of the drug treatments of interest (cyclosporine A, eltrombopag, romiplostin, danazol, or methenolone) during the follow-up period and before the first transfusion record, if any.

SUMMARY:
This was a retrospective non-interventional cohort study with secondary use of data from the Medical Data Vision (MDV) hospital-based database to evaluate the effectiveness of early drug intervention in preventing transfusion compared to watchful observation among adult transfusion-independent aplastic anemia (AA) patients in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Having at least one confirmed diagnosis of AA within the selection period (1 inpatient or 2 outpatient claims per the International Statistical Classification of Diseases, 10th Revision [ICD-10] code, without any suspicion flag).
* Being aged 15 to 90 years at the index date.
* Having at least 3 months of continuous enrolment prior to the index date.

Exclusion Criteria:

* Having a blood transfusion recorded any time before the index date.
* Having anti-thymocyte globulin (ATG) treatment recorded within 3 months after the index date.
* Having at least one prescription record for any of the drug treatments of interest any time before the index date.
* Having a diagnosis of acute myeloid leukemia (AML), chronic myelomonocytic leukemia (CMML) or other leukemia any time before the index date.
* Having an AA diagnosis (without suspicious flag) date earlier than the start of patient's observation in the database.
* Having less than 6 months of continuous follow-up.

Safety Population - Additional Exclusion Criterion:

- Having a diagnosis of hepatotoxicity, kidney dysfunction, hypertension, or diabetes mellitus any time before the index date.

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 1603 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Probability of Having Blood Transfusion in the Matched Effectiveness Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Crude Hazard Ratios of Having Blood Transfusion After 6 Months of Follow-up in the Matched Effectiveness Population | Baseline, 6 months
Adjusted Hazard Ratios of Having Blood Transfusion After 6 Months of Follow-up in the Matched Effectiveness Population | 6 months

SECONDARY OUTCOMES:
Sex | Baseline
Age | Baseline
Weight | Baseline
Body Mass Index (BMI) | Baseline
Number of Patients With Aplastic Anemia, per Severity Level | Baseline
Number of Patients With Immune Thrombocytopenia (ITP) Diagnosis Before Index Date | Baseline
Number of Patients With Myelodysplastic Syndrome (MDS) Diagnosis Before Index Date | Baseline
Number of Patients With Pre-index Comorbidities | Baseline
Number of Patients With Pre-index Use of Chloramphenicol | Baseline
Platelet Count | Baseline
Neutrophil Count | Baseline
Hemoglobin Level | Baseline
Number of Patients Per Treatment Therapy in the Matched Effectiveness Population | Baseline
Number of Patients With Aplastic Anemia in the Matched Effectiveness Population, per Severity Level | Baseline
Number of Patients in the Matched Effectiveness Population Who Discontinued | Baseline, at 6 and 9 months, and at 1 and 2 years
Probability of Having Blood Transfusion in Early Drug Intervention and Watchful Observation Matched Patients From the Effectiveness Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having Stem-Cell Transplantation (SCT) in Early Drug Intervention and Watchful Observation Matched Patients From the Effectiveness Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having Anti-Thymocyte Globulin (ATG) in Early Drug Intervention and Watchful Observation Matched Patients From the Effectiveness Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having Blood Transfusion at Different Timepoints by Drug Categories in the Matched Effectiveness Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having SCT at Different Timepoints by Drug Categories in the Matched Effectiveness Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having ATG at Different Timepoints by Drug Categories in the Matched Effectiveness Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having a Bleeding Event in Early Drug Intervention and Watchful Observation Matched Patients From the Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having Cataract in Early Drug Intervention and Watchful Observation Matched Patients From the Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having Diabetes in Early Drug Intervention and Watchful Observation Matched Patients From the Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having Hepatotoxicity in Early Drug Intervention and Watchful Observation Matched Patients From the Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having Hypertension in Early Drug Intervention and Watchful Observation Matched Patients From the Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having an Infection in Early Drug Intervention and Watchful Observation Matched Patients From the Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having Kidney Dysfunction in Early Drug Intervention and Watchful Observation Matched Patients From the Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having Acute Myeloid Leukemia (AML), Chronic Myelomonocytic Leukemia (CMML) or Another Leukemia in Early Drug Intervention and Watchful Observation Matched Patients From the Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having MDS in Early Drug Intervention and Watchful Observation Matched Patients From the Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having Paroxysmal Nocturnal Hemoglobinuria (PNH) in Early Drug Intervention and Watchful Observation Matched Patients From the Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having a Thromboembolic Event in Early Drug Intervention and Watchful Observation Matched Patients From the Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having Myelofibrosis in Early Drug Intervention and Watchful Observation Matched Patients From the Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having a Bleeding Event by Drug Categories in the Matched Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having Cataract by Drug Categories in the Matched Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having Diabetes by Drug Categories in the Matched Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having Hepatotoxicity by Drug Categories in the Matched Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having an Infection by Drug Categories in the Matched Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having Kidney Dysfunction by Drug Categories in the Matched Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having AML, CMML or Another Leukemia by Drug Categories in the Matched Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having MDS by Drug Categories in the Matched Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having PNH by Drug Categories in the Matched Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having a Thromboembolic Event by Drug Categories in the Matched Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.
Probability of Having Myelofibrosis by Drug Categories in the Matched Safety Population | Baseline, at 6 and 9 months, and at 1, 2, 5, and 10 years
  The Kaplan-Meier survival analysis technique was used to estimate probability.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, Tokyo, Japan